CLINICAL TRIAL: NCT00762333
Title: Circulating Markers for Ischemic Heart Disease
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Bruce Liang, Professor of Medicine, Director Pat and Jim Calhoun Cardiovascular Center, UConn Health
Other Study IDs: 07-252-2; 59806
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Ischemia; Congestive Heart Failure
MeSH Terms: conditions — Myocardial Infarction; Ischemia; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Myocardial Infarction

SUMMARY:
The purpose of this research is to determine if two proteins in the blood are increased during acute myocardial infarction and whether their levels are higher in those who develop heart failure than those who do not. These two proteins are produced and potentially released when the heart muscle is damaged. They may then be released into the blood and be detected by standard method in the research laboratory. At this time, detection of an increase in these proteins in the blood is not known to be associated with any disease or myocardial infarction.

DETAILED DESCRIPTION:
Hypotheses, Objectives and Aims:

Hypotheses:Caspase-3, cleaved and activated, and dystrophin can be detected in human circulation. The levels of these two markers are elevated during acute myocardial infarction. Furthermore, the levels of these two proteins are greater in those who develop heart failure than those who do not.

Objectives:

* To determine whether cleaved caspase-3 and dystrophin can be detected in human circulation after an acute myocardial infarction
* To compare serum levels of these two markers in those who develop heart failure and those who do not

Scientific Background and Significance: Apoptosis is a regulated biological process resulting in cell death (4-9). Caspases, a family of cysteine acid proteases regulate the process, and in fact, lead to apoptosis. Apoptotic trigger or signal results in the activation of proximal or initiator caspases (such caspase-8, -9, 10). These initiator caspases then cleave and in turn activate downstream effector caspases such as caspases-3, -6 and -7. These effector caspases then cleave various proteins such as those present in cytoskeletons and nucleus like lamin A, alpha-fodrin and poly (ADP-ribose) polymerase, leading to apoptosis. Caspase-3 is the key executioner in this apoptotic pathway, responsible totally or critically in the proteolytic cleavage of cellular and nuclear proteins. Activation of caspase-3 requires proteolytic processing of its inactive zymogen into active p17 and p12 fragments. The cleaved caspase-3 can be detected by antibodies specific for this cleaved enzyme (p17 fragment) in cell lysates by immunoblotting or by an ELISA assay utilizing spectrophotometric determination with a microplate reader at OD450 nm. Ischemia and reperfusion are known to cause apoptosis. Therefore, acute MI may be associated with release of the final executioner of apoptosis that is caspase-3, into the circulation.Another potential marker for acute deterioration is dystrophin. Dystrophin was originally identified as the x-linked gene whose mutations in its N-terminus cause cardiomyopathy. Dystrophin provides important structural support for the cardiac myocyte and its sarcolemmal membrane (10-11). It links actin at its N-terminus with the dystrophin-associated protein complex and sarcolemma at the C-terminus and the extracellular matrix of muscle. Mutations cause loss of support and sarcolemmal instability and myopathy. Myocardial dystrophin translocation and cleavage are associated with the progression of heart failure and contractile dysfunction. These changes are reversed following reduction of mechanical stress from ventricular assistance device (12). Since MI is associated with sarcolemmal instability, dystrophin may also be released into circulation.

ELIGIBILITY:
Inclusion Criteria:

* men and women, 18 years of age and over with acute myocardial infarction (determined by positive cardiac markers -CKMB/ troponin) with or without heart failure (dyspnea, rales, edema, elevated jugular venous pressure, ascites).
* Heart failure can be diagnosed using imaging evidence such as dilated heart, poor contractile function or echocardiographic Doppler evidence of diastolic dysfunction or elevated right- or left-sided filling pressures
* A control group of male subjects age 60 and older without history of MI or heart disease

Exclusion Criteria:

* Subjects unable to give consent
* Subjects who have undergone cardiac or non-cardiac surgery in the 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are two arms to this study:
  The investigators hope to enroll 350 healthy individuals, as defined by having no prior diagnosis of heart disease to determine baseline levels and diurnal variations of the markers.
  Participants being evaluated for an acute Myocardial Infarction as determined by positive CK MB/troponin levels, will be asked to enroll.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2007-06; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for acute myocardial infarction, stroke or death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T. Liang, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States